CLINICAL TRIAL: NCT06336616
Title: Getting Out of the House: A Behavioral Activation Approach to Support Community Participation With Individuals With Serious Mental Illness
Brief Title: Getting Out of the House: Using Behavioral Activation to Increase Community Participation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 31164
Record Dates: First submitted 2024-02-27; First posted 2024-03-29 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Major Depressive Disorder; Schizo Affective Disorder; Schizophrenia; Bipolar Disorder
Keywords: serious mental illness
MeSH Terms: conditions — Depressive Disorder, Major; Psychotic Disorders; Schizophrenia; Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): All participants will receive an online behavioral intervention for 10 weeks, followed by monthly maintenance sessions for 3 months.
  Interventions: Behavioral: Behavior Activation

INTERVENTIONS:
Behavioral: Behavior Activation — Participants will be taught to identify meaningful activities, set goals, use environmental cues, self-reward, to identify barriers and facilitators, and learn new skills to support them to develop self-management skills and new habits.
  Other Names: SWITCH

SUMMARY:
The goal of this study is to evaluate the effectiveness of an behavioral activation intervention to increase meaningful activity and community participation for people with serious mental illness.

The overall objective of this study is to increase engagement in meaningful activities and community participation. The objectives of the project are as follows:

1. To determine if the intervention leads to increases the frequency and variety of activities.
2. To determine if the intervention leads to increases in community mobility.
3. To determine which demographic and environmental factors and mechanisms of action impact the effectiveness of the intervention.
4. To determine if the the intervention leads to an improvement in overall well-being (e.g., improved quality of life).

Participants will be asked to attend a 2-hour weekly online session for 10 weeks and then a 1-hour online monthly session for a 3 month maintenance period.

For data collection, participants will also be asked to:

1. Complete three, approximately 1-hour interviews at baseline, after the 10 week intervention, and again at the end of the maintenance period;
2. Carry a mobile phone with a global positioning system app to track their movements outside their home for 2 weeks at a time, at three separate times (e.g., baseline, after the intervention, and at the end of the maintenance period); and
3. Complete a 15 minute weekly interviews for 26 weeks about their daily activities and participation.

The study will enroll 52 participants split into 4 cohorts of 13. The study will use a multiple baseline design and, as such, all participants will receive the intervention and there is no control group.

ELIGIBILITY:
Inclusion Criteria:

1. must respond yes to three questions related to their history with serious mental illness (see below);
2. a score of 8 or higher on the Center for Epidemiologic Studies Depression Scale - Revised -10 (CES-D-R-10)
3. have Internet access;
4. be willing to carry a cell phone with a GPS tracking application;
5. indicate that they would like to participate more in the community;
6. be able to communicate in English;
7. be over the age of 18; and
8. and be available on for the day and time (i.e., Monday, Tuesday, Wednesday, Thursday, or Friday) the intervention is scheduled for each cohort.

Questions related to history with serious mental illness:

1. "Have you ever been told by a psychiatrist or other mental health professional that you have major depression, bipolar disorder, manic depression, schizophrenia or schizoaffective disorder?",
2. "Have you ever been hospitalized for this mental health or emotional problem?", and
3. "Has this mental health or emotional problem substantially interfered with or limited your ability to participate in any major life activities such as work, school, recreation, social activities, religious activities, family relationships, or caring for yourself?" Answering yes to these 3 questions would be indicative of a lifetime serious mental illness.

Exclusion Criteria:

1. those who are unable to give informed consent
2. those who report having a legal guardian -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Activity Logs | administered 26 times: 1 time per week for 26 weeks.
  The activity logs are open ended forms in which participants are asked to enter in the primary activities they did in a day (e.g., work), the amount of time they did if for (e.g., 2 hours), how effortful it was on a scale of 1-5, and what their mood was before, during, and after the activity on a scale of 1-5. A higher score on effort (5) is indicative of greater effort, and a higher score ono mood indicates a better or more positive mood. Activities type will be analyzed qualitatively.
Participation Checklist | administered 26 times: 1 time per week for 26 weeks
  Participants will be asked to state whether they did an activity from a list of 20 items. Response options include yes or no. A greater number of "yes" responses will indicate a greater level of participation that week.
Behavior Activation for Depression Scale | administered 26 times: 1 time per week for 26 weeks
  The behavior activation depression scale measures related to activity, social interaction, and negative thinking or feelings There are 25 statements measured on a 6-point Likert scale varying from not at all to completely. The range of scores is 0 to 54, with high scores representing higher behavioral activation.activities
Temple University Community Participation Measure | administered 3 times: at baseline, within 1 month following the 10 weeks of weekly meetings, and 3 months later within 1 month following the intervention
  Measures engagement in 29 participation areas, if those areas are important to them, how often they did them and if it was enough, not enough, or too much. Higher reported frequency across a greater number of areas indicates higher rates of participation. Higher number of activities reported as being important and done enough indicate greater sufficiency of participation.
Community Mobility (Global Positioning System; GPS) | administered 3 times for 2 weeks: at baseline, within 1 month following the 10 weeks of weekly meetings, and 3 months later within 1 month following the end of the intervention
  Participants will carry a cellphone that will track their movements in the community using a GPS app. GPS data shows movements in the community in distance traveled in kilometers. This will be analyzed as total distance traveled.
Community Mobility (Global Positioning System; GPS) | administered 3 times for 2 weeks: at baseline, within 1 month following the 10 weeks of weekly meetings, and 3 months later within 1 month following the end of the intervention
  Participants will carry a cellphone that will track their movements in the community using a GPS app. GPS data shows locations participants go to in the community with GPS coordinates. This will be analyzed as the number of locations visited.

SECONDARY OUTCOMES:
Lerman Quality of Life Interview | administered 3 times: at baseline, within 1 month following 10 week intervention, and within 1 month following the maintenance period 3 months later
  This measure assesses the overall perceived quality of life. There are 11 items across three domains: community inclusion, holistic health and functioning, and human and legal rights. The statement "[If homeless or in jail, the place where you typically sleep at night?]" will be removed from Q5 the questionnaire as it is not relevant to our study participants. Response options vary from terrible to delighted on a 7-point scale. Responses closer to 7 (delighted) indicate greater perceived quality of life and responses closer to 1 (terrible) indicate lower perceived quality of life. The scores will be summed across questions and higher scores indicate better perceived quality of life.
New General Self-Efficacy Scale (adapted to participation) | administered 3 times: at baseline, within 1 month following the 10 week intervention, and within 1 month following the maintenance period 3 months later
  This is a self-report measure of self-efficacy or perceived ability to participate in the community. There are 10 items with 4 responses options ranging from not at all (1) to exactly true (4). Total scores can range from 10-40 with a higher score indicated greater self-efficacy
Recovery Assessment Scale (RAS) | administered 3 times: at baseline, within 1 month following the 10 week intervention, and within 1 month following the maintenance period 3 months later
  Three subscale from the RAS will be used: 1) reliance on others, 2) confidence and hope, and 3) willingness to ask for help. Responses range from strongly disagree (1) to strongly agree (5). Scores can range from 16-80 with higher scores indicating greater recovery, reliance on others, confidence, and willingness to ask for help.
Activity Assessment Scale | administered 3 times: at baseline, within 1 month following 10 week intervention, and within 1 month following the maintenance period 3 months later
  Measures motivation, ease, pleasure, and satisfaction related to behaviors that are precursors to participation (e.g., planning transportation and outings). Each subscale (e.g., motivation) is measured on a 4-point scale from "not at all" to "extremely." Each subscale is scored separately with scores ranging from 5 to 20. Higher scores indicate higher level of each subscale (e.g. ease).
Capabilities and Opportunities for Participation Questionnaire | administered 3 times: at baseline, within 1 month following the 10 week intervention, and within 1 month following the maintenance period 3 months later
  Includes 8 statements related to capabilities tied to participation (e.g., I feel comfortable taking public transportation) and 14 related to opportunities tied to participation (e.g., I have access to materials or equipment to participate). All items are measure on a scale of 1-6 from strongly disagree to strongly agree. For 17 of the 22 items higher scores indicate greater capabilities and opportunities and for 5 of the 22 lower scores indicate greater capabilities and opportunities.
Self-Control and Self-Management Scale | administered 3 times: at baseline, within 1 month following the 10 week intervention, and within 1 month following the maintenance period 3 months later
  The 16-item instrument includes statements about self-control and self-management. The scoring is on a 6-point Likert scale, and the anchors adopted for score reporting are 1 to 6. Thus, the possible total scale score range is 16-96 with higher scores indicating greater self-management and self-control.
Habit Strength Scale | administered 3 times: at baseline, within 1 month following the 10 week intervention, and within 1 month following the maintenance period 3 months later
  This was modified to measures habit strength for participation rather than moderate to vigorous activity. The measure consists of 17 items or statements with response options ranging from 1-6 on a 6-point Likert scale from strongly disagree to strongly agree. Possible scores range from 17 to 102 with higher scores indicating greater habit strength.
University of California Los Angeles Loneliness Scale | administered 3 times: at baseline, within 1 month following the 10 week intervention, and within 1 month following the maintenance period 3 months later
  These 3 questions are only being given to people who report having a mental illness. The questions related to how often people feel socially isolated or lonely. Response options range from 1) hardly ever, 2) some of the time, and 3) often. Responses (3) indicate increased loneliness and more "hardly ever" responses indicate less loneliness.
Lehman Quality of LIfe (QOL) Interview Social Relations sub scale | administered 3 times: at baseline, within 1 month following the 10 week intervention, and within 1 month following the maintenance period 3 months later
  This subscale is an indicator of social relationships and networks. It contains 6-items rated on a 5-point scale and 6 additional measures on a 7-point scale. Higher scores on the items indicate better social relationships.
Hopkins Symptoms Checklist | administered 3 times: at baseline, within 1 month following the 10 week intervention, and within 1 month following the maintenance period 3 months later
  This measure assesses primary symptom dimensions over the past week using a 25-item assessment with a 4-point Likert scale (0 = not at all to 4 = extremely). Higher scores indicate higher levels of symptoms. Separate averages of depression and anxiety items are calculated and a total score represents the mean of the total 25 items.
The Life Engagement Test | administered 3 times: at baseline, within 1 month following the 10 week intervention, and within 1 month following the maintenance period 3 months later
  The measure assesses purpose in life. There are 6 items/statements with response options on a 5-point Likert scale ranging from 1-5, (1= "Strongly disagree" and 5 = "Strongly agree"). Scores for each question are summed with a range of scores from 6 to 30. Higher scores indicate greater levels of purpose in life.
The University of Rhode Island Change Assessment Measure (URICA) | administered 3 times: at baseline, within 1 month following the 10 week intervention, and within 1 month following the maintenance period 3 months later
  The measure contains 28 items with statements related to readiness to change. The readiness score is determined by calculating the means for precontemplation, contemplation, action, and the maintenance responses. The mean from the precontemplation is then subtracted from the summation of the means of the other three stages. 8 or lower classified as people in Precontemplation, 8-11 classified as people in Contemplation, and 11-14 classified as people in Preparation or Action.
Reward Probability Index | administered 3 times: at baseline, within 1 month following the 10 week intervention, and within 1 month following the maintenance period 3 months later
  The 20-item self-report measure designed assess the likelihood of environmental rewards. Each question is scored on a scale of 1-4 from strongly disagree to strongly agree. Higher scores on 11 of the 20 items and lower scores on 9 of the items indicate a greater likelihood of environmental reward.

CONTACTS AND LOCATIONS:
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States